CLINICAL TRIAL: NCT04146389
Title: Hyperprolactinemia and Adrenal Steroidogenesis: is There a Link?
Brief Title: Hyperprolactinemia and Adrenal Steroidogenesis
Acronym: Prado
Status: Terminated | Type: Observational
Why Stopped: Preliminary analyses of the samples provide no indication for a clinically relevant relationship between hyperprolactinemia and stimulation of adrenal steroidogenesis.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Prado
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Hyperprolactinemia
Keywords: adrenal steroidogenesis; doping
MeSH Terms: conditions — Hyperprolactinemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore the effects of prolactin on adrenal steroid profiles in patients with hyperprolactinemia due to prolactinomas before and after initialisation of treatment.

DETAILED DESCRIPTION:
Prolactin is known to influence many biological processes. One potential target is the adrenal gland, where prolactin may stimulate the production of adrenal steroid hormones. Conditions of increased prolactin production(hyperprolactinemia) could, therefore, increase concentrations of adrenal steroids. One of the potential implications would be false doping accusations of athletes engaging in elite sports.

This interaction between prolactin and adrenal steroidogenesis, however, remains poorly understood, and the available research findings are conflicting.

The investigators, therefore, seek to explore the relationship between prolactin and adrenal steroidogenesis by monitoring prolactin levels and blood and urinary steroid profiles of patients with hyperprolactinemia due to prolactinomas before and after treatment initialisation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Female and pre-menopausal
* Serum prolactin > 150 ng/ml

Exclusion Criteria:

* Corticotropic and/or thyreotropic insufficiency
* Pregnancy, planned pregnancy or breastfeeding
* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Incapacity to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve up to 17 pre-menopausal female individuals with hyperprolactinemia due to prolactinomas, who will undergo treatment at the University Hospital Bern.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Covariation of plasma prolactin and plasma dehydroepiandrosterone | From pre-treatment till 5 weeks of treatment
  Covariation of plasma prolactin and plasma dehydroepiandrosterone over time

SECONDARY OUTCOMES:
Change in the plasma steroid profile | From pre-treatment till 5 weeks of treatment
  Change in the plasma steroid profile over time
Change in plasma prolactin levels | From pre-treatment till 5 weeks of treatment
  Change in plasma prolactin levels over time
Change in the urine steroid profile | From pre-treatment till 5 weeks of treatment
  Change in the urine steroid profile over time
Covariation of urinary adrenal steroids | From pre-treatment till 5 weeks of treatment
  Covariation of urinary adrenal steroids over time

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Inselspital, Bern University Hospital, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland